CLINICAL TRIAL: NCT02395445
Title: A Comparison of Tracheal Intubation Using the Totaltrack vs the Macintosh Laryngoscope in Routine Airway Management: a Randomised, Controlled Clinical Trial
Brief Title: A Comparison of Tracheal Intubation Using the Totaltrack vs the Macintosh Laryngoscope in Routine Airway Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manuel Ángel Gómez-Ríos (Other)
Responsible Party: Sponsor-Investigator, Manuel Ángel Gómez-Ríos, M.D., Complexo Hospitalario Universitario de A Coruña
Organization: Complexo Hospitalario Universitario de A Coruña (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MGR-TT-2015-F1
Record Dates: First submitted 2015-03-09; First posted 2015-03-23 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Endotracheal Intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Totaltrack (Active Comparator): Indirect laryngoscopy
  Interventions: Device: orotracheal intubation
- Macintosh Laryngoscope (Active Comparator): Direct laryngoscopy
  Interventions: Device: orotracheal intubation

INTERVENTIONS:
Device: orotracheal intubation

SUMMARY:
Endotracheal intubation is usually required to allow unrestricted surgical approach. The Macintosh laryngoscope is the standard method. However in certain situations as difficult airway this technique is ineffective and poorly tolerated by the patient. Fiberoptic intubation is the gold standard in this scenario, however sometimes it is not possible due to failure or unavailability, so alternatives are needed. The TotalTrack (MedComflow SA, Barcelona, Spain) has been designed specifically for the airway management. However, despite its use in clinical practice, there are no comparative studies regarding direct laryngoscopy

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective general anesthesia requiring OTI.
* Patients duly informed and they have signed the informed consent during the pre-anesthetic consultation, or be sought after due meditation, expressing its consent to the inclusion in the study.
* Age ≥18 years.
* ASA I-III.
* Sufficient intellectual capacity to understand the procedure and equipment used.
* Do not submit predictors of difficult airway (Mallampati class III or IV; thyromental distance <6 cm, sternomental distance <12.5 cm, interincisal distance<4.0 cm, bite test II or III, cervical mobility <90 ° or history of difficult intubation).
* Do not undergo thyroid surgery or present pharyngolaryngeal, glottic or cervical pathology
* BMI <30kg / m2
* Not presenting risk factors for aspiration
* Not presenting respiratory disease, coronary or cerebral vascular.
* Do not have a sore throat preoperative

Exclusion Criteria:

* Failure to meet the above criteria
* Pregnancy
* Allergy to any drug included in the protocol.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2015-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Total time of successful intubation with the Macintosh laryngoscope and TotalTrack. | Time of Orotracheal intubation (TOTI) (up to 1 hour)

SECONDARY OUTCOMES:
IDS Scale | TOTI (up to 1 hour)
POGO Score | TOTI (up to 1 hour)
number of maneuvers | TOTI (up to 1 hour)
Number of attempts of endotracheal intubation | TOTI (up to 1 hour)
Position taken by the anesthesiologist during orotracheal intubation | TOTI (up to 1 hour)
hemodynamic response | OTI pre and postintubation (up to 10 minutes)
  Heart Ratio, Arterial Pressure
Complications | OTI and postintubation ( up to 24 hours)
endotracheal intubation success rate of each device | TOTI (up to 1 hour)
Degree of satisfaction | time of postintubation (up to 10 minutes)
  Visual Analogic Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Manuel Ángel Gómez-Ríos, A Coruña, A Coruña, Spain

REFERENCES:
- [Background] Pearce A. Evaluation of the airway and preparation for difficulty. Best Pract Res Clin Anaesthesiol. 2005 Dec;19(4):559-79. doi: 10.1016/j.bpa.2005.07.004. PMID 16408534
- [Background] Adnet F, Borron SW, Racine SX, Clemessy JL, Fournier JL, Plaisance P, Lapandry C. The intubation difficulty scale (IDS): proposal and evaluation of a new score characterizing the complexity of endotracheal intubation. Anesthesiology. 1997 Dec;87(6):1290-7. doi: 10.1097/00000542-199712000-00005. PMID 9416711
- [Background] Ochroch EA, Hollander JE, Kush S, Shofer FS, Levitan RM. Assessment of laryngeal view: percentage of glottic opening score vs Cormack and Lehane grading. Can J Anaesth. 1999 Oct;46(10):987-90. doi: 10.1007/BF03013137. PMID 10522589